CLINICAL TRIAL: NCT00552825
Title: Pulmonary Function at Presentation and Follow-up in Hemato-Oncology 3-7 Years
Brief Title: Pulmonary Function at Presentation and Follow-up in Hemato-Oncology 3-7 Years Old Children
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Other Study IDs: SHEBA-05-3889-OE-CTIL; Observational
Record Dates: First submitted 2007-11-01; First posted 2007-11-02 (Estimated); Last update posted 2007-11-02 (Estimated); Status verified 2007-11

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloblastic Leukemia; Solid Tumors,; Hodgkin's Disease; Non-Malignant
Keywords: acute lymphoblastic leukemia; long-term lung function
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: all were in a single group

SUMMARY:
The aim of this study was to investigate the occurrences of respiratory symptoms risk factors and abnormalities in lung function in young children (3-6 years old) with hemato-oncologic diseases at presentation (before treatment) and up to 3 years follow-up (study period).

DETAILED DESCRIPTION:
Pulmonary function tests (PFTs) are a part of the routine follow-up of patients receiving anti-cancer treatment. Treatment is frequently associated with diverse pulmonary damage which may become functionally and clinically evident many years later. PFTs may help to quantify the damage in the lungs; help to evaluate the point at which lung function deviates from normal to allow early intervention before irreversible lung damage occurs and thereby to reduce morbidity and mortality.

Reliable PFTs in the preschool age have traditionally been difficult to perform, but recent publications have demonstrated that the majority of preschool children can produce reproducible forced expiratory flow volume (FEVC) curves with proper coaching techniques. This recent development may enable studying the long term effect (years) of treatment on lung function in young children suffering from hemato-oncologic diseases.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric patients (age 3-7 years) with hemato-onclogic diseases that were treated at the Hemato-Oncology Department, and were sent to the pediatric pulmonary unit.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All pediatric patients (age 3-7 years) with hemato-onclogic diseases that were treated at the Hemato-Oncology Department, and were sent to the pediatric pulmonary unit at the Safra children's hospital, Sheba medical center, Ramat-Gan, Israel, to perform lung function tests, as a part of a 3-year follow-up study.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2005-10; Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ori Efrati, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical CenterPediatric pulmonary unit, Pulmonary function laboratory, Ramat Gan, Ramat Gan, Israel